CLINICAL TRIAL: NCT04683900
Title: Mediterranean Diet Intervention to Improve Gastrointestinal Function in Parkinson's Disease: a Randomized, Controlled, Clinical Trial
Brief Title: Mediterranean Diet Intervention to Improve Gastrointestinal Function in Parkinson's Disease a Randomized, Controlled, Clinical Trial
Acronym: MEDI-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB202001333
Record Dates: First submitted 2020-12-17; First posted 2020-12-24 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Parkinson Disease
Keywords: Mediterranean diet; Microbiome; Constipation; Inflammation
MeSH Terms: conditions — Parkinson Disease; Constipation; Inflammation | interventions — Standard of Care; Diet, Mediterranean; Methods

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, controlled parallel study in which participants either follow a Mediterranean diet or their habitual diet for an 8-week intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care + Mediterranean Diet (Experimental): Participants will be given standard of care for constipation (handout) plus individualized diet education on the Mediterranean diet and instructed to follow the diet during the 8-week intervention period. Diet education will be administered by a study dietitian and followed with weekly phone calls to ensure compliance, improve adherence to the diet and monitor for adverse events.
  Interventions: Other: Standard of care + Mediterranean diet (intervention)
- Standard of Care (Active Comparator): Participants will be given standard of care for constipation (handout) to utilize during the 8-week intervention period. A study dietitian will follow up with weekly phone calls to support adherence and monitor for adverse events.
  Interventions: Other: Standard of care (control)

INTERVENTIONS:
Other: Standard of care + Mediterranean diet (intervention) — Participants will receive a constipation management handout that is distributed regularly to patients who present with constipation symptoms at an outpatient neurology clinic. The handout recommends increasing fluids daily, as well as increasing physical activity and dietary fiber intake. Laxative medications and recommendations for usage are included.
  Participants will be instructed to include the following in their diet: a) abundant use of olive oil for cooking and dressing dishes; b) consume ≥2 daily servings of vegetables; c) ≥2-3 daily serving of fruits; d) ≥3 weekly servings of legumes; e) ≥3 weekly servings of fish/seafood; f) ≥3 weekly serving of nuts/seeds; g) select white instead of red or processed meats; h) cook at least twice a week with sofrito. Limit consumption of cream, butter, processed meat, sugared beverages, industrial bakery products and desserts, and French fries or chips. For usual drinkers, the main source of alcohol should be wine.
  Arms: Standard of Care + Mediterranean Diet
Other: Standard of care (control) — Participants will receive a constipation management handout that is distributed regularly to patients who present with constipation symptoms at an outpatient neurology clinic. The handout recommends increasing fluids daily, as well as increasing physical activity and dietary fiber intake. Laxative medications and recommendations for usage are included.
  Arms: Standard of Care

SUMMARY:
This is a 10-week randomized, controlled study to investigate the effect of a Mediterranean diet intervention on gastrointestinal function in Parkinson's disease. After a 2-week run-in period, participants will be instructed to receive standard of care for constipation or receive standard of care + follow a Mediterranean diet for 8 weeks and answer daily and weekly questionnaires. Nutritional and neurological evaluations and stool samples will be collected at 0, 4 and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed Parkinson's disease aged 40-85 years
* Drug naïve or on stable dosage of Parkinson's medications with no plans to change for the duration of the study protocol
* Hoehn & Yahr stage =<2.5 in the clinical "ON" state
* Constipation syndrome scores >=2.0 based on the GSRS
* Consume <20 grams of fiber daily based on the Block Fruit/Vegetable/Fiber screener
* Able to complete informed consent in English
* Willing to maintain habitual diet through the pre-baseline period.
* Willing to make dietary changes to follow a Mediterranean diet and/or receive standard of care for constipation during the intervention period.
* Willing to complete daily and weekly questionnaires and 12 dietary recalls over approximately 10 weeks.
* Able to provide stool samples during the study collection periods.
* Willing to avoid strenuous exercise and alcohol such as beer, wine, and cocktails 24 hours prior to each of the 3 study visits.
* Able to fast (no food or drink, except water, or decaf tea) at least 12 hours before each study visit
* Willing to discontinue taking prebiotic, herbal, or high-dose vitamin or mineral supplements that may impact inflammation during the pre-baseline period and throughout the study protocol.

Exclusion Criteria:

* Atypical or secondary Parkinsonism
* Underweight (BMI <18.5)
* History of deep brain stimulation (DBS) surgery
* Regular use of enemas or suppositories to alleviate constipation (e.g., >1 time per week)
* Use of another investigational product within 3 months of the screening visit
* Antibiotic or probiotic supplement use within 2 months from the day of stool collection
* Currently being treated for a physician-diagnosed GI disease or condition other than constipation, irritable bowel disease, gastroparesis, reflux or diverticular disease

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
GSRS Constipation Syndrome Score | 10 weeks
  The difference between mean change (final - baseline) in constipation syndrome scores for the Med diet versus control diet.

SECONDARY OUTCOMES:
Stool Frequency | Each week up to 10 weeks
  Compare the number of stools between the intervention and control groups
Stool Form | Each day up to 10 weeks
  Compare stool form, as measured by the Bristol Stool Form Scale (BSFS), between the intervention and control groups. The BSFS is scored between 1 (hard stool) - 7 (liquid stool).
Laxative Usage | Each week up to 10 weeks
  Compare number of days using laxative medications between the intervention and control groups.
Digestive Health | Every week up to 10 weeks
  Weekly GI symptoms assessed using the Gastrointestinal Symptom Rating Scale (GSRS). The GSRS consists of 15 questions related to 5 syndromes, constipation, diarrhea, reflux, abdominal pain, and indigestion. Symptoms are scored 1=no discomfort to 7=very severe discomfort. Scores from each of the 15 questions are summed for the total GSRS score.
Quality of Life Related to Digestive Health | Every week up to 10 weeks
  Weekly GI experiences assessed using an in-house Digestion-Associated Quality of Life questionnaire.
Fecal Microbial Diversity | Baseline (Week 0); Midpoint (Week 4); Final (Week 8)
  Changes in fecal microbial composition and diversity (i.e. alpha and beta diversity) will be assessed.
Fecal Microbial Quantitative Polymerase Chain Reaction (qPCR) | Baseline (Week 0); Midpoint (Week 4); Final (Week 8)
  Changes in fecal microbial composition to quantify bacterial species of interest (e.g., F. prausnitzii, Prevotella, Roseburia, Bilophila, Akkermansia, etc.) will be assessed.
Intestinal Inflammation and Permeability | Baseline (Week 0); Midpoint (Week 4); Final (Week 8)
  Changes in fecal calprotectin and zonulin will be assessed using enzyme-linked immunosorbent assay

OTHER OUTCOMES:
Mediterranean diet adherence | Each week up to 10 weeks
  Compare Mediterranean diet adherence scores using the 14-Item Mediterranean diet adherence screener (MEDAS) between groups
Dietary Fiber Intake | Baseline (Week 0); Midpoint (Week 4); Final (Week 8)
  Changes in dietary fiber intake as measured by averaged 4-day dietary recalls using the Automated Self-Administered 24-hour dietary recall (ASA-24) between groups
Body weight | Baseline (Week 0); Midpoint (Week 4); Final (Week 8)
  Changes in body weight between groups
Body Composition (Fat Free Mass) | Baseline (Week 0); Midpoint (Week 4); Final (Week 8)
  Changes in fat free mass using bio-impedance spectroscopy (BIS) between groups
Handgrip strength | Baseline (Week 0); Midpoint (Week 4); Final (Week 8)
  Changes in handgrip strength will be assessed using a hand dynamometer between groups
Quality of Life (QOL) | Baseline (Week 0); Midpoint (Week 4); Final (Week 8)
  Changes in QOL will be assessed using the Parkinson's Disease Quality of life -39 (PDQ-39)
Anxiety | Baseline (Week 0); Midpoint (Week 4); Final (Week 8)
  Changes in symptoms of anxiety will be assessed using the Hamilton Anxiety Rating Scale
Depression | Baseline (Week 0); Midpoint (Week 4); Final (Week 8)
  Changes in symptoms of anxiety will be assessed using the Hamilton Depression Rating Scale
Physical Activity | Baseline (Week 0); Midpoint (Week 4); Final (Week 8)
  Changes in MET minutes will be assessed using the International Physical Activity Questionnaire (IPAQ).

CONTACTS AND LOCATIONS:
Overall Officials: Bobbi Langkamp-Henken, PhD, RD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The anonymized datasets used and/or analyzed during the study will be available from the corresponding author upon reasonable request and approval of the University of Florida.

REFERENCES:
- [Derived] Rusch C, Beke M, Tucciarone L, Dixon K, Nieves C Jr, Mai V, Stiep T, Tholanikunnel T, Ramirez-Zamora A, Hess CW, Langkamp-Henken B. Effect of a Mediterranean diet intervention on gastrointestinal function in Parkinson's disease (the MEDI-PD study): study protocol for a randomised controlled trial. BMJ Open. 2021 Sep 22;11(9):e053336. doi: 10.1136/bmjopen-2021-053336. PMID 34551955